CLINICAL TRIAL: NCT05156983
Title: A Phase 3, Prospective, Randomized, Open-label, Adaptive Group Sequential, Multicenter Trial With Blinded Endpoint Assessment to Evaluate the Efficacy and Safety of TAK-330 for the Reversal of Direct Oral Factor Xa Inhibitor-induced Anticoagulation in Patients Requiring Urgent Surgery/Invasive Procedure
Brief Title: A Study of TAK-330 to Reverse the Effects of Factor Xa Inhibitors For Adults Needing Urgent Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAK-330-3001; 2021-004138-12 (EudraCT Number); 2022-503012-16-00 (EU CTIS Number: EU CTIS)
Record Dates: First submitted 2021-12-13; First posted 2021-12-14 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Coagulation Disorder
Keywords: Reversal of Factor Xa inhibitors
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Intervention Model Description: Adaptive parallel-group sequential design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAK-330 25 IU/kg (Experimental): Participants will receive TAK-330, 25 international unit per kilogram (IU/kg) single intravenous infusion on Day 1 (prior to surgery) as an initial dose and an additional dose of 25 IU/kg TAK-330 can be administered during the surgery if deemed necessary by the surgeon. The total dose of TAK-330 administered to the participant should not exceed 50 IU/kg or 5,000 IU, whichever is smaller.
  Interventions: Drug: TAK-330
- SOC 4F-PCC (Active Comparator): Participants will receive 4F-PCC (excluding Prothromplex Total and activated 4F-PCC) as standard of care (SOC) on Day 1 (prior to surgery). The dose and infusion speed of the SOC 4F-PCC will be based on local institutional protocols. An additional dose of SOC 4F-PCC not exceeding total dose of 50 IU/kg or 5,000 IU, whichever is smaller can be given during the surgery if required.
  Interventions: Drug: SOC 4F-PCC

INTERVENTIONS:
Drug: TAK-330 — Participants will receive TAK-330, 25 IU/kg single intravenous infusion on Day 1 and an additional dose of 25 IU/kg TAK-330 can be administered if required.
  Arms: TAK-330 25 IU/kg
Drug: SOC 4F-PCC — Participants will receive 4F-PCC as SOC on Day 1. The dose and infusion speed of the SOC 4F-PCC will be based on local institutional protocols. An additional dose of SOC 4F-PCC not exceeding total dose of 50 IU/kg or 5,000 IU, whichever is smaller can be given during the surgery if required.
  Arms: SOC 4F-PCC

SUMMARY:
The aim of this study is to find out the effects of TAK-330 compared with four-factor prothrombin complex concentrate (4F-PCC) as part of standard treatment other than Prothromplex Total for anticoagulation reversal in participants treated with Factor Xa inhibitors who require urgent surgery/invasive procedure.

The participant will be assigned by chance to either TAK-330 or SOC 4F-PCC as part of standard treatment before surgery.

Patients participating in this study will need to be hospitalized. They will also be contacted (via telehealth/phone call) 30 days after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participant or legally authorized representative willing to sign e-consent/written informed consent form.
* Participants at least 18 years of age at enrollment.
* Participant currently on treatment with oral Factor Xa inhibitor (rivaroxaban, apixaban, edoxaban).
* In the opinion of the surgeon, the participant requires an urgent surgery/procedure that is associated with high-risk of intraoperative bleeding within 15 hours from the last dose of Factor Xa inhibitor and requires a reversal agent for suspected direct oral Factor Xa inhibitor-related coagulopathy. For participants who are beyond the 15-hour window, eligibility requires proof of elevated plasma anti-Factor Xa (FXa) levels using either specific direct oral anti-coagulant (DOAC)-calibrated (apixaban, rivaroxaban or edoxaban) anti-FXa levels of greater than (>) 75 nanograms per milliliter (ng/mL), or heparin calibrated anti-FXa assay levels of >0.5 international unit per milliliter (IU/mL) at screening.
* Women of childbearing potential should have a negative pregnancy test documented prior to enrollment.

Exclusion Criteria:

* The participant has an expected survival of less than 30 days, even with best available medical and surgical care.
* Recent history (within 90 days prior to screening) of venous thromboembolism, myocardial infarction (MI), disseminated intravascular coagulation (DIC), ischemic stroke, transient ischemic attack, hospitalization for unstable angina pectoris or severe or critical coronavirus 2 (SARS-CoV-2) infection.
* Active major bleeding defined as bleeding that requires surgery or transfusion of >2 units of packed red blood cell (PRBC) or intracranial hemorrhage with the exception of subacute and chronic subdural hemorrhages with a Glasgow Coma Score (GCS) greater than or equal to (>=) 9.
* Polytrauma for which reversal of Factor Xa-inhibition alone would not be sufficient to achieve hemostasis.
* Known prothrombotic disorder including primary antiphospholipid syndrome, antithrombin-3 deficiency, homozygous protein C deficiency, homozygous protein S deficiency, and homozygous factor V Leiden.
* Known bleeding disorder (example, platelet function disorders, hemophilia, Von Willebrand disease, or coagulation factor deficiency).
* Platelet count less than (<) 50,000 per microliter (/mcL).
* History of heparin-induced thrombocytopenia.
* Administration of procoagulant drugs (example, non-study prothrombin complex concentrates (PCCs), recombinant Factor VIIa) or blood products (transfusion of whole blood, fresh frozen plasma, cryoglobulins, plasma fractions, or platelets) within 7 days before enrollment. (Note: administration of PRBCs for hemoglobin correction, tranexamic acid or aminocaproic acid are not exclusion criteria).
* Planned use of procoagulant drugs (example, Vitamin K, non-study PCCs, recombinant Factor VIIa) or blood products (transfusion of whole blood, fresh frozen plasma, cryoglobulins, plasma fractions, or platelets) after enrollment but before the 24±4 hours hemostatic assessment (Key secondary endpoint). Planned administration of tranexamic acid (TXA) or aminocaproic acid after randomization but before the start of IP infusion, should be noted during randomization to properly stratify these participants in the interactive response technology (IRT). Planned administration of TXA or aminocaproic acid after start of IP infusion but before the 24±4 hours hemostatic assessment is prohibited. Administration of any of the above products before the 24±4 hours hemostatic assessment will impact the assessment of hemostasis. Administration of PRBCs for hemoglobin correction, is not an exclusion criterion.
* Administration of unfractionated heparin within 2 hours before randomization or low molecular weight heparin within 6 hours before randomization.
* Hypersensitivity to PCC constituents or any excipient of TAK-330.
* Participants with history of confirmed immunoglobulin A (IgA) deficiency with hypersensitivity reaction and antibodies to IgA.
* Septic shock as defined by persistent hypotension requiring vasopressors to maintain mean arterial pressure (MAP) >=65 millimeters of mercury (mmHg) and having blood lactate >2 millimole (mmol) despite adequate volume resuscitation.
* Acute or chronic liver failure (hepatic cirrhosis Child-PUGH score C)
* Renal failure requiring dialysis
* Any other condition that could, in the opinion of the investigator, put the participant at undue risk of harm if the participant were to participate in the study.
* Participation in another clinical study involving an investigational product or device within 30 days prior to study enrollment, or planned participation in another clinical study involving an investigational product or device during the course of this study. Participation in an observational study is not an exclusion criterion.
* The use of PROTHROMPLEX TOTAL as SOC 4F-PCC.
* Women who are breastfeeding at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2028-04-12 (Estimated); Study Completion 2028-04-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Intraoperative Effective Hemostasis | At the end of the surgery/procedure
  Percentage of participants achieving intraoperative effective hemostasis, as determined by the Intraoperative Four Point Hemostatic Efficacy Scale and assessed by the principal investigator (PI), the surgeon, or a qualified member of the surgical team.

SECONDARY OUTCOMES:
Percentage of Participants With Postoperative Effective Hemostasis | At 24 hours after the end of investigational product infusion
  Percentage of participants achieving postoperative effective hemostasis at 24±4 hours following the completion of investigational product infusion, as determined by the Postoperative Four Point Hemostatic Efficacy Scale and assessed by the PI, the surgeon, or a qualified member of the surgical team.
Percentage of Participants With Intraoperative Effective Hemostasis Based on Hemostatic Efficacy Rating Algorithm | At the end of the surgery/procedure
  Percentage of participants achieving intraoperative effective hemostasis, as determined by the Hemostatic Efficacy Rating Algorithm and assessed by the PI, the surgeon, or a qualified member of the surgical team.
Number of Participants With Usage of Blood Products or Non-Study Hemostatic Agents for Bleeding Control | Within 24 hours after the end of investigational product infusion
  Number of participants with usage of blood products or non-study hemostatic agents for bleeding control will be documented from the end of IP infusion to 24 hours after end of study product infusion.
Number of Units of Packed Red Blood Cells (PRBCs) Administered to Achieve Bleeding Control | Within 24 hours after the end of investigational product infusion
  Number of units of PRBCs administered to achieve bleeding control within 24 hours after the end of IP infusion.
Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interests (AESIs) | Within 30 days after the end of the surgery/invasive procedure (up to 33 days)
  An Adverse Event (AE) is defined as any untoward medical occurrence (including a symptom or disease or an abnormal laboratory finding) in a participant or clinical investigation participants administered a medicinal product and which does not necessarily have a causal relationship with the treatment. TEAEs are defined as those with a start date on or after the first dose of study treatment, or with a start date before the date of first dose of study treatment but increasing in severity after the first dose of study treatment. A SAE is any event that results in: death; life-threatening event; requires inpatient hospitalization or results in prolongation of existing hospitalization; persistent or significant disability/incapacity; results in a congenital anomaly/birth defect or a medically important event. AESI will include hypersensitivity reactions, events of disordered coagulation such as bleeding and hypercoagulability.
Number of Participants With Thrombotic Events | Within 30 days after the end of the surgery/invasive procedure (up to 33 days)
  Number of thrombotic events within 30 days after the end of the surgery/invasive procedure will be assessed. Thrombotic events occur when a blood clot, known as a thrombus, is formed within a blood vessel. It prevents blood from flowing normally through the circulatory system.
Number of Participants With Deaths Within 30 Days Post-Surgery/Invasive Procedure | Within 30 days post-surgery/invasive procedure (up to 33 days)
  Number of deaths Within 30 days post-surgery/invasive procedure will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (63):
- United States (13):
  - University of Arkansas Medical Sciences, Arkansas City, Arkansas
  - University of California Davis Health System, Sacramento, California
  - Denver Metro Orthopedics, P.C., Englewood, Colorado
  - University of Florida, Gainesville, Florida
  - Rutgers, The State University of New Jersey, New Brunswick, New Jersey
  - ECU Health Medical Center, Greenville, North Carolina
  - Metro Health Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Ascension St. John Medical Center, Tulsa, Oklahoma
  - University of Pennsylvania - Perelman School of Medicine, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Carilion Medical Center, Virginia Beach, Virginia
- Argentina (4):
  - Hospital Universitario Austral, Buenos Aires
  - Clinica Zabala, Ciudad Autonoma Buenos Aires
  - Fundacion para la Lucha contra las Enfermedades Neurologicas de la Infancia - FLENI, Ciudad Autonoma Buenos Aires
  - Hospital Privado de Rosario, Santa Fe
- Austria (2):
  - LKH - Universitaetsklinikum Graz, Graz
  - Landesklinikum Neunkirchen, Neunkirchen
- Belgium (4):
  - ZOL, Genk, Limburg
  - Jessa Ziekenhuis Hospital, Hasselt, Limburg
  - AZ Groeninge, Kortrijk
  - CHU UCL Namur, Therasse 1
- Brazil (3):
  - Irmandade da Santa Casa da Misericordia de Santos, Santos, São Paulo
  - Hospital de Clinicas de Ijui, Ijuí
  - Hospital Sao Paulo, São Paulo
- Canada (6):
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre (LHSC) - University Hospital, London, Ontario
  - Unity Health Toronto St Michaels Hospital, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - The Ottawa Hospital - General Campus, Ontario
  - CHU de Quebec- Hopital de l Enfant Jesus, Québec
- Czechia (3):
  - Fakultni nemocnice Brno, Jihlavska
  - Fakultni nemocnice v Motole, Prague (Praha)
  - Dept of II. interni klinika - gastroenterologie, Srobarova C
- France (5):
  - CHU Strasbourg - Hopital Hautepierre, Strasbourg, Bas Rhin
  - Hospital michallon - CHUGA, Grenoble
  - Hopital Marie Lannelongue, Le Plessis-Robinson
  - Hôpital Lariboisière, Paris
  - GH Paris Saint Joseph, Paris
- Germany (4):
  - BG Klinikum Murnau gGmbH, Murnau am Staffelsee, Bavaria
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden, Saxony
  - Universitaetsklinikum Leipzig AoeR, Leipzig, Saxony
  - Klinikum Dortmund gGmbH, Murnau am Staffelsee
- Konstantopoulio General Hospital, N.Ionia, Nea Ionia, Attica, Greece
- Hungary (4):
  - Bekes Varmegyei Kozponti Korhaz, Békéscsaba, Attica
  - Ozdi Almasi Balogh Pal Korhaz, Szeged, Attica
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem, Debrecen
- Israel (8):
  - Shamir Medical Center (Assaf Harofe), Beer Yaacov
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Rabin MC, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Uniwersytecki Szpital Kliniczny nr 1 im. prof. Tadeusza Sokołowskiego PUM w Szczecinie, Szczecin, Poland
- Portugal (2):
  - Centro Hospitalar do Baixo Vouga, E.P.E. - Unidade de Aveiro, Aveiro
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E, Rua Conceição Fernandes
- Spain (3):
  - Hospital Clinico Universitario de Salamanca, Salamnca, Salamanca
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/61ba5ab5f571d4002a64b4aa